CLINICAL TRIAL: NCT02788799
Title: Clinical Impact of Pre-hospital Posterior ECG Leads Implementation for Identifying Occlusion of Left Circumflex Coronary Artery in ST Segment Elevation Myocardial Infarction
Brief Title: Finding LCX AMI With Posterior ECG LeadS
Acronym: FLAWLESs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Nykøbing Falster County Hospital (Other); Region Sjælland (Other)
Responsible Party: Principal Investigator, Yama Fakhri, MD, Rigshospitalet, Denmark
Other Study IDs: FLAWLESS-16-YF
Record Dates: First submitted 2016-05-26; First posted 2016-06-02 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Myocardial Infarction
Keywords: ST Elevation; LCX Artery
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

GROUPS / COHORTS (2):
- Control
  Interventions: Other: Standard 12-Lead ECG
- Intervention
  Interventions: Other: Standard 12-Lead ECG; Other: Posterior ECG Leads

INTERVENTIONS:
Other: Standard 12-Lead ECG — Conventional record of Standard 12-lead ECG in every patient with suspect of acute coronary syndrome.
Other: Posterior ECG Leads — Recording posterior ECG leads (V7, V8 and V9) in addition to standard 12-lead ECG for identifying STEMI involving left cirumflex coronary artery.
  Other Names: Posterior Leads (V7, V8 and V9)
  Groups: Intervention

SUMMARY:
Along with symptoms of chest pain, the presence of ST segment elevations on ECG is the criterion usually used in practice to identify patients with acute coronary artery occlusion and is essential for the direct and acute referral of patients for primary PCI. However, ECG does not always reflect changes in the posterior wall of the heart, often equivalent to the left circumflex coronary artery's (LCX) supply area, resulting in an underrepresentation of LCX as culprit artery in STEMI populations. There is a general concern that some patients with genuine acute occlusion of LCX may present without ST segment elevation and be denied reperfusion therapy, resulting in larger infarction and worse outcome.

The aim of this trial is to implement record of posterior ECG leads (V7, V8 and V9) in addition to the standard 12-lead ECG in the pre-hospital setting and to evaluate the clinical impact of this implementation: In comparison to a control cohort of STEMI patients diagnosed with a pre-hospital standard 12-lead ECG prior study start, the investigators hypothesize that introducing V7-V9 leads as a clinical routine in the pre-hospital setting will identify patients with STEMI involving LCX and with a non-diagnostic standard 12-lead ECG.

ELIGIBILITY:
Inclusion Criteria: Intervention group:

* All STEMI patients referred directly from the pre-hospital setting, treated with primary PCI and with available standard 12-lead ECG and ECG with V7-V9 leads.

Exclusion Criteria:

* STEMI patients treated with primary PCI and no ECG with V7-V9 leads.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The intervention group will contain STEMI patients referred directly from the pre-hospital setting to PCI-center for primary PCI during study periode. In these patients, both standard 12-lead ECG and ECG with V7-V9 leads will be recorded and tele-transmitted to the PCI-center.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with LCX occlusion as culprit artery in the intervention group compared to the control group | Day one - culprit lesion treated with primary PCI

SECONDARY OUTCOMES:
Proportion of patients in the intervention group with STEMI involving LCX artery, non-diagnostic standard 12-lead ECG and ST segment elevation >0,5 mm in ≥2 leads in posterior ECG leads (V7-V9). | Day one - culprit lesion treated with primary PCI

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kastrup, MD,Professor, Study Chair — Dept of Cardiology, Rigshospitalet, Copenhagen, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark